CLINICAL TRIAL: NCT02482012
Title: Minor Increase Over Minimal Risk Without Direct Patient Benefit Research in the NICU: Parental and Staff Perspectives
Brief Title: Minor Increase Over Minimal Risk Research in NICU
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: CCC#34099
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Infant, Premature; Infant, Late; Infant, Preterm; Infant
Keywords: research; vulnerable population; 45 CFR 46.406
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Staff: Staff nurses and physicians in the NICU
  Interventions: Other: Survey
- Parents: Parents of infants in the NICU and a smaller group of parents of infants in the well baby nursery.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — This was a survey

SUMMARY:
Infants comprise a potentially vulnerable research population that received special consideration and protections under the US Code of Federal Regulations - Subpart D. Of the four categories of research involving children, 45 CFR 46.406 is of particular interest to researchers, ethicists, parents, and clinical staff members since it concerns the conduct of research with "more than minimal risk" without the prospect of direct benefit. Parents are the surrogate decision makers for infants. When asked about this type of research in studies pertaining to older infants and children, parent themes include: concerns of medical research and research-related risk, desire to advance generalizable medical knowledge and knowledge specific to their own child's disease. There are no data on parents' perceptions regarding this category of research that target the premature, late-preterm and term newborn populations.

This study involves a questionnaire for both staff (nurses and physicians) and parents. The questionnaire represented 4 different infant scenarios in a random order. Respondents are asked to answer questions related to enrollment in a research study for each of the 4 scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants in the NICU
* Parents of infants on well-baby nursery
* NICU Staff (nurses and physicians)

Exclusion Criteria:

* Non-English Speaking
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NICU staff and parents of infants
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
determination of willingness to participate in research | 15 minutes
  This is a survey to determine attitudes / willingness to participate in a specific category of research.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Locke, DO, MPH, Principal Investigator — Christiana Care Health Services, Inc.
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States